CLINICAL TRIAL: NCT06345079
Title: A Randomised Study of Cessation of Somatostatin Analogues After Peptide Receptor Radionuclide Therapy in Mid, Hind-Gut and Pancreatic Neuroendocrine Tumours (STOPNET)
Brief Title: Cessation of Somatostatin Analogues After PRRT in Mid, Hind-Gut and Pancreatic Neuroendocrine Tumours
Acronym: STOPNET
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Australasian Gastro-Intestinal Trials Group (Network)
Collaborators: Canadian Cancer Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AG0219NET
Record Dates: First submitted 2024-03-14; First posted 2024-04-03 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Neuroendocrine Tumors
Keywords: Advanced; Unresectable grade 1 or 2; mid, hind- gut or pancreatic neuroendocrine tumours
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continue SSA (Active Comparator): Patients randomised to continue SSA will receive a SSA injection ≥28 days prior to the first PRRT cycle, during PRRT cycle, and every 4 weeks after completion of PRRT.
  Interventions: Drug: Continuation of somatostatin analogues
- Cease SSA (Experimental): Patients randomised to cease SSA will receive SSA injection ≥28 days prior to their first cycle of PRRT. Patients will not receive any further long acting SSA injections after this time.
  Interventions: Drug: Cessation of somatostatin analogues

INTERVENTIONS:
Drug: Cessation of somatostatin analogues — Patients randomised to cease SSA will receive their last SSA injection ≥28 days prior to their first cycle of PRRT and will remain off SSA for the duration of the study. If there is concern from the treating team that a patient may experience a carcinoid flare after PRRT, then short acting octreotide is allowed to be used to control any symptoms.
  Other Names: SSA cessation
  Arms: Cease SSA
Drug: Continuation of somatostatin analogues — Patients randomised to continue SSA will receive a SSA injection ≥28 days prior to their first cycle of PRRT, during PRRT and will continue receiving SSA every 4 weeks after PRRT.
  Other Names: SSA continuation
  Arms: Continue SSA

SUMMARY:
Neuroendocrine tumours (NETs) are slow growing cancers, which commonly present as metastatic incurable disease. Some neuroendocrine tumours, termed functional NETs, overproduce hormones which result in a variety of symptoms. However, approximately 75% of NETs are considered non-functional meaning that they do not result in hormone overproduction. The main treatment for both functional and non-functional NETs is somatostatin analogues (SSA, a type of inhibitory hormone). These drugs slow tumour growth and reduce hormone production. Over time, the majority of patients will experience tumour growth despite treatment with SSA therapy. When this occurs, the addition of Peptide Receptor Radionuclide Therapy (PRRT, a type of targeted radiotherapy) in combination with ongoing SSA therapy is given. However, it is not known if continuing SSA therapy after commencement of PRRT is beneficial or not.

The aim of this study is to estimate the outcomes of patients with grade 1 and 2 well differentiated mid, hind-gut or pancreatic neuroendocrine tumours who have progressed on SSA therapy and receive subsequent PRRT with or without concurrent SSA.

DETAILED DESCRIPTION:
Neuroendocrine tumours commonly originate from the gut and metastasise widely including to the liver, lymph nodes and bones. Originally called "carcinoid tumours", these cancers are most commonly treated with somatostatin analogues (SSA) first line. These analogues treat carcinoid syndrome and slow tumour growth. Despite SSA therapy, progression develops over time. Upon progression, peptide receptor radionuclide therapy (PRRT) is the next standard therapeutic option. After PRRT is initiated, it is unclear if continuing SSA injections is beneficial. There are reasons to believe it might be necessary to continue SSAs, but other reasons to believe they should cease. Given that SSA injections are expensive and associated with side effects, this study aims to clarify the utility of continuing SSA injections after progression on SSA therapy and commencement of PRRT.

STOPNET aims to explore outcomes in grade 1 and 2 mid, hind gut or pancreatic neuroendocrine tumours, that have progressed on SSA therapy, are eligible to receive PRRT and in whom the SSA is either continued or ceased after PRRT is commenced.

The two primary objectives include

1. To estimate the 20-month progression free survival rate after PRRT commencement in patients who cease and who continue SSA.
2. Feasibility as measured by:

   1. Recruitment rate and
   2. Patient acceptance of ceasing and staying off SSA over the 20 month follow up period.

The study design of STOPNET is prospective, randomised, non-comparative, open label, multicentre phase II study. Patients meeting the inclusion and exclusion criteria will be randomised, prior to commencing PRRT, to either continue or cease SSA treatment. Randomisation will occur centrally in REDCap by the AGITG STOPNET study team. Randomisation will be 2:1 (the majority being randomised to cease SSA) and will be stratified by WHO tumour grade (1 V 2), sites of metastases (visceral only verse visceral and bone) and institution.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years of age with well or moderately differentiated mid or hindgut neuroendocrine tumour, or pancreatic neuroendocrine tumour, metastatic and inoperable, demonstrating progression despite SSA treatment of sufficient disease magnitude to warrant PRRT as determined by the treating clinician and/or the NET Multidisciplinary Team (MDT).
* Must have measurable disease on triphasic CT/MRI as per RECIST 1.1.
* Ki67 ≤ 20% AND mitotic count 20 per HPF (i.e., WHO grade 1 or 2)
* Patient has been receiving growth-controlling doses of SSA for at least 12 weeks prior to study entry. This is a minimum of 30 mg Octreotide or120mg lanreotide monthly.
* Uptake on SSTR PET scan demonstrating somatostatin receptor expression that is suitable for PRRT as judged by the clinical team. FDG PET scans are to be done at the judgement of the treating team and are not required for enrolment into this study.
* PRRT is deemed the most appropriate next treatment step (i.e., patient is inoperable, and liver directed therapies are not preferred)
* ECOG performance status 0 -2
* Written informed consent. Patients must be willing to either cease or continue SSA, depending on which study arm they are randomised to. Patients must be willing to comply with all other study requirements
* Adequate renal, hepatic and haematologic function as judged by the treating team
* Life expectancy of at least 12 months
* Availability of tissue from resection or biopsy samples is desired but is not mandatory for study inclusion. Tissues will only be retrieved if the patient consents to optional translational research sample collection. Similarly, bloods for research purposes will only be collected from those patients who consent to optional translational research sample collection.
* Non-functioning NET: SSA treatment will have been commenced for control of tumour growth and not for carcinoid or other hormone overproduction syndrome, as judged by the clinician and/or NET MDT. Non-functioning NET is judged by the treating clinical team based on patient symptomatology. In addition, for this study, non-functioning tumour is defined as:

  * 24-hour urine 5-hydroxyindoleacetic acid (5HIAA) of <1.5x upper limit of normal (applies to mid and hind gut patients only).
  * Please note: routine measurement of gastrin, insulin, C-peptide levels, glucagon etc. is not required unless clinically indicated.
  * Never had escalation of the SSA treatment dose to control carcinoid carcinoid or other hormone-related symptoms
  * Never required short acting SSA treatment to control carcinoid carcinoid or other hormone-related symptoms
  * No significant carcinoid induced valvular heart disease IE: Echocardiogram to be done in all patients within 26 weeks of study enrolment and deemed safe to proceed with PRRT by the treating team.

Exclusion Criteria:

* This study is for pancreatic, mid-gut and hind-gut NET only. Gastric and lung NETs are excluded
* Any patient on an SSA dose lower than the standard growth-control dose. Patients must have been on octreotide 30 mg or lanreotide 120 mg for at least 3 months prior to study entry.
* Prior chemotherapy or targeted therapy (e.g., everolimus). Patients who have received prior local therapy, including external beam radiotherapy and liver directed therapy prior to or during SSA therapy are eligible.
* Any contraindication to PRRT, as per local institutional practice.
* Pregnancy. For female patients of childbearing potential and male patients with a female partner who is of childbearing potential, contraception and counselling is required.
* Prior PRRT. Patients being considered for re-treatment with PRRT are not eligible
* Uncontrolled central nervous system metastases. Patients must have completed any surgery or radiation at least 4 weeks prior to registration and must be off corticosteroids for at least 2 weeks
* Any patient, in the opinion of the investigator, who will not comply with study assessments and follow up visits. These might include any social, psychological, or geographical concerns, including alcohol/drug abuse
* Any poorly controlled concurrent medical illness that may prevent the patient from complying with study assessments and follow up. This is to be judged by the treating team
* Any concurrent or prior malignancy that, in the opinion of the treating team, may interfere with study assessments and endpoints

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
20-month progression free survival rate after PRRT | 20 months
  Estimate the 20-month progression free survival rate after PRRT in patients who cease and who continue SSA.
Assess the barriers which would impede the feasibility of a subsequent phase 3 trial | 20 months
  1. Proportion of participants that remained on the SSA cessation arm for the duration of the 20-month study follow up (patient acceptance of SSA cessation).
  2. Rate of recruitment: ability to complete recruitment over the 24-month recruitment period

SECONDARY OUTCOMES:
Measure Quality of life using the European Organisation For Research And Treatment Of Cancer (EORTC) Core Quality of Life questionnaire (QLQ-C30) scales | 20 months
  Responses to the QLQ-C30 scale from 0-100 using EORTC guidelines, with higher scores reflecting better level of functioning.
Measure Quality of life using the EORTC QLQ-GINET21 scales | 20 months
  Responses to the QLQ-GINET21 scale from 0-100 using EORTC guidelines, with higher scores reflecting more severe symptoms.
Cost-effectiveness of SSA therapy cessation | The MBS/PBS data will be obtained for the period six months prior to study entry, and until the end of 2 years follow-up post PRRT for patients who have provided consent.
  Access to Medicare and PBS data to asses use of other healthcare providers, diagnostic tests and imaging services funded via public health care systems and use of pharmaceutical services respectively.
Psycho-oncological impacts of SSA therapy cessation: Decision Regret | 20 months
  Psycho-oncological impacts of SSA therapy cessation using the self-reported measures of Decision Regret Scale from 1 - 5 (1-Strongly Agree, 2-Agree, 3-Neither Agree Nor Disagree, 4-Disagree, 5-Strongly Disagree)
Psycho-oncological impacts of SSA therapy cessation: Fear of Cancer Progression | 20 months
  Psycho-oncological impacts of SSA therapy cessation using the self-reported measures of the Fear of Cancer Progression Scale from 1 - 5 (1-Never, 2-Seldom, 3-Sometimes, 4-Often, 5-Very often)
Psycho-oncological impacts of SSA therapy cessation: Decisional Conflict | 20 months
  Psycho-oncological impacts of SSA therapy cessation using the self-reported measures of the Decisional Conflict Scale from 0 - 4 (0-Strongly Agree, 1-Agree, 2-Neither Agree Nor Disagree, 3-Disagree, 4-Strongly Disagree)
Time to commencement of subsequent therapy | 20 months
  Time to commencement of subsequent therapy (e.g re-challenge with PRRT, liver directed therapies, chemotherapy, targeted therapies)
Overall survival | 20 months
  Estimate the 20-month overall survival rate in patients who cease and who continue SSA.
Rates of SSA being recommenced over time | 20 months
  Cumulative percentage of SSA recommencement over time.

OTHER OUTCOMES:
Exploratory analyses | 20 months
  Exploratory analyses including, but not limited to: Define and validate NET tissue and circulating biomarkers with a particular focus on miRNA.

CONTACTS AND LOCATIONS:
Locations (12):
- Australia (6):
  - Royal North Shore Hospital, Sydney, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Royal Brisbane and Womens Hospital, Brisbane, Queensland
  - The Queen Elizabeth Hospital, Adelaide, South Australia
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Fiona Stanley Hospital, Perth, Western Australia
- Canada (6):
  - BC Cancer Agency, Vancouver Cancer Centre, Vancouver, British Columbia
  - London Health Sciences Centre Research Institute (LHSCRI), London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Odette Cancer Centre Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No